CLINICAL TRIAL: NCT05132569
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Tolebrutinib (SAR442168) in Adults With Generalized Myasthenia Gravis (MG)
Brief Title: Efficacy and Safety of Tolebrutinib (SAR442168) Tablets in Adult Participants With Generalized Myasthenia Gravis
Acronym: URSA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: For strategic reasons the Tolebrutinib MG study has been terminated
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC17262; U1111-1265-6378 (Registry Identifier: ICTRP); 2021-003898-59 (EudraCT Number)
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Results first posted 2024-04-08 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo/Tolebrutinib (Placebo Comparator): Participants with moderate-to-severe gMG received placebo (matched to tolebrutinib) tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period. Participants who completed the DB period entered the OLE period and received tolebrutinib 60 milligrams (mg) orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
  Interventions: Drug: Tolebrutininb; Drug: Placebo
- Tolebrutinib/Tolebrutinib (Experimental): Participants with moderate-to-severe gMG received tolebrutinib 60 mg tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period. Participants who completed the DB period entered the OLE period and continued to receive tolebrutinib 60 mg orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
  Interventions: Drug: Tolebrutininb

INTERVENTIONS:
Drug: Tolebrutininb — Pharmaceutical form: Film-coated tablet Route of administration: Oral
Drug: Placebo — Pharmaceutical form: Film-coated tablet Route of administration: Oral
  Arms: Placebo/Tolebrutinib

SUMMARY:
This was a multicenter, randomized, double-blind, placebo-controlled, Phase 3 study to evaluate the efficacy and safety of tolebrutinib compared with placebo in adult participants aged 18 to 85 years old with moderate-to-severe generalized myasthenia gravis (gMG), who received Standard of Care (SoC). The double-blind (DB) treatment period of 26 weeks comprised of 7 site visits followed by a 2-year open label extension (OLE) period with quarterly visits. The efficacy of tolebrutinib versus placebo during the DB period was assessed by clinical evaluations, including scales based on physician examination or direct participant feedback i.e., patient reported outcomes (PROs). These evaluations continued during the OLE to measure long term efficacy and safety.

DETAILED DESCRIPTION:
The duration of the DB period was 26 weeks. The OLE was planned up to 104 weeks. The duration of the whole study DB+OLE was planned up to130 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants were 18 years of age to 85 years of age inclusive, at the time of signing the informed consent.
* Participants with a diagnosis of gMG at screening with generalized muscle weakness meeting the clinical criteria for diagnosis of MG, as defined by the myasthenia gravis foundation of America (MGFA) Clinical Classification Class II, III, or IV, and likely not in need of a respirator for the duration of the study, as judged by the Investigator.
* Positive serologic testing for anti-acetylcholine receptor (anti-AChR) or anti-muscle-specific kinase (anti-MuSK) autoantibody at screening OR
* Seronegative for both anti-AChR and anti-MuSK autoantibodies and with prior diagnosis supported by greater than or equal to (>=) 1 of the following 3 tests:

  1. History of abnormal neuromuscular transmission demonstrated by single-fiber electromyography or repetitive nerve stimulation.
  2. History of positive edrophonium chloride test.
  3. Participant had demonstrated improvement in gMG signs on oral acetylcholinesterase inhibitors as assessed by the treating physician.
* The participant had a total score >=6 on myasthenia gravis-activities of daily living scale at screening and Day 1 with greater than half of the score attributed to non-ocular items.

Exclusion Criteria:

* MGFA Class I (ocular MG) or Class V.
* Participants had undergone thymectomy within 6 months of screening or having a planned thymectomy during the trial period.
* The participant had a history of infection or might be at risk for infection: A history of active or latent tuberculosis (TB); Participants at risk of developing or having reactivation of hepatitis; Persistent chronic or active recurring infection required treatment with antibiotics, antivirals, or antifungals; Fever within 4 weeks of the Screening Visit (>=38 degree Celsius; however, if due to brief and mild ear, nose, throat viral infection participant might be included based on the Investigator's judgment); A history of infection with human immunodeficiency virus (HIV); A history of T-lymphocyte or T-lymphocyte-receptor vaccination, transplantation (including solid organ, stem cell, and bone marrow transplantation) and/or antirejection therapy.
* Any malignancy within the past 5 years prior Screening Visit (except for effectively treated carcinoma in situ of the cervix, adequately treated non-metastatic squamous or basal cell carcinoma of the skin and malignant thymoma that had been resected or were considered as cured by any treatment with no evidence of metastatic disease for >=3 years) will be exclusionary.
* Conditions that might predispose the participant to excessive bleeding.
* Clinically significant laboratory abnormalities (including evidence of liver injury) or electrocardiogram abnormalities at Screening.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- United States (5):
  - Georgetown University-Site Number:8400008, Washington D.C., District of Columbia
  - SFM Clinical Research, LLC-Site Number:8400006, Boca Raton, Florida
  - University of South Florida Health- Morsani Center for Advanced Healthcare-Site Number:8400001, Tampa, Florida
  - Harvard Medical School - Brigham and Women's Hospital-Site Number:8400004, Boston, Massachusetts
  - Neurology Center of San Antonio, PA-Site Number:8400009, San Antonio, Texas
- Canada (2):
  - Investigational Site Number :1240004, Edmonton, Alberta
  - Investigational Site Number :1240003, London, Ontario
- China (3):
  - Investigational Site Number :1560003, Chengdu
  - Investigational Site Number :1560001, Shanghai
  - Investigational Site Number :1560002, Wuhan
- Hungary (2):
  - Investigational Site Number :3480002, Pécs
  - Investigational Site Number :3480001, Szeged
- Italy (4):
  - Investigational Site Number :3800002, Milan, Lombardy
  - Investigational Site Number :3800001, Milan
  - Investigational Site Number :3800004, Napoli
  - Investigational Site Number :3800003, Roma
- Investigational Site Number :3920002, Sagamihara-shi, Kanagawa, Japan
- Investigational Site Number :6160001, Zabrze, Poland
- Spain (2):
  - Investigational Site Number :7240003, L'Hospitalet de Llobregat, Catalunya [Cataluña]
  - Investigational Site Number :7240005, Madrid, Madrid, Comunidad de
- United Kingdom (2):
  - Investigational Site Number :8260002, Exeter, Devon
  - Investigational Site Number :8260001, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: EFC17262 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25263&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 22 sites in 9 countries from 03-Dec-2021 to 21-Feb-2023. A total of 6 participants were randomized in a 1:1 ratio to receive treatment with tolebrutinib or placebo.
Pre-assignment Details: Randomization was stratified by Myasthenia Gravis Foundation of America (MGFA) class (II, IIIa/IVa, or IIIb/IVb) and region (United States [US], non-US). Due to early termination of the study by sponsor, several planned efficacy analysis were not performed for the study.
Groups:
- Placebo/Tolebrutinib: Participants with moderate-to-severe generalized myasthenia gravis (gMG) received placebo (matched to tolebrutinib) tablet orally once daily as an add-on therapy to their Standard of Care (SoC) for 26 weeks in the double-blind (DB) treatment period. Participants who completed DB period entered the open label extension (OLE) period and received tolebrutinib 60 milligrams (mg) orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
- Tolebrutinib/Tolebrutinib: Participants with moderate-to-severe gMG received tolebrutinib 60 mg tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period. Participants who completed DB period entered the OLE period and continued to receive tolebrutinib 60 mg orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
Period: DB Period: 26 Weeks
Arm/Group | Placebo/Tolebrutinib | Tolebrutinib/Tolebrutinib
Started | 3 | 3
Completed | 2 | 1
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Study terminated by sponsor | 1 | 1
Period: OLE: Week 27 Till Termination (Week 61)
Arm/Group | Placebo/Tolebrutinib | Tolebrutinib/Tolebrutinib
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Study terminated by sponsor | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants. Based on the low enrolment number and in order to protect and maintain participant privacy/confidentiality, data were reported under a single arm.
Groups:
- Overall Participants: Participants with moderate-to-severe gMG received tolebrutinib 60 mg tablet or matched placebo tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period. Participants who received treatment with tolebrutinib 60 mg orally daily in the DB period entered the OLE period and continued the same treatment in the OLE period. Participants who received matched placebo in the DB period received tolebrutinib 60 mg orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
Arm/Group | Overall Participants
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Change From Baseline in Myasthenia Gravis-activities of Daily Living (MG-ADL) Total Score at Week 26
Description: The MG-ADL is an 8-item patient-reported categorical scale that assesses MG symptoms and their effects on daily activities. The MG-ADL targeted symptoms and disability across ocular (2 items), bulbar (3 items), respiratory (1 items), and gross motor or limb impairment (2 items) symptoms. It evaluates a participant's capacity to perform different activities in their daily life. Each item is scored on a 4-point scale ranged from 0 (normal) to 3 (severe), where higher score represents the more severe symptoms or impaired performance. MG-ADL total score is the sum of each item score which ranged from 0 (normal) to 24 (severe). Higher score represents severe disability due to MG. DB period Baseline value was defined as last available value prior to the first dose of the study medication in the DB period.
Time Frame: Baseline (Day 1), Week 26
Population: Evaluable data was collected for 3 participants only; and thus, was not presented to protect participant confidentiality.
Groups:
- DB Period: Placebo: Participants with moderate-to-severe gMG received placebo (matched to tolebrutinib) tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period.
- DB Period: Tolebrutinib: Participants with moderate-to-severe gMG received tolebrutinib 60 mg tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period.
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: OLE Period: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events Leading to Permanent Study Intervention Discontinuation and Adverse Events of Special Interests (AESIs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. A SAE was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was a medically important event. An AESI was defined as one of scientific & medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was considered appropriate. Relatedness to study vaccine was based on Investigator's discretion.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: Analysis was performed on the safety population which included all randomized participants who took at least 1 dose of study intervention and were analyzed according to the intervention they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- OLE Period: Placebo/Tolebrutinib: Participants who completed the DB period entered the open label extension (OLE) period and received tolebrutinib 60 mg orally once daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
- OLE Period: Tolebrutinib/Tolebrutinib: Participants who completed the DB period entered the OLE period and continued to receive tolebrutinib 60 mg orally once daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 2 | 1
Participants
  AEs | 2 | 0
  SAEs | 0 | 0
  AEs leading to permanent study intervention discontinuation | 0 | 0
  AESIs | 0 | 0

3. Primary Outcome: OLE Period: Number of Participants With Hematological Abnormalities
Description: Hematological parameters assessed were: platelet count, red blood cell count, hemoglobin, hematocrit, white blood cell, neutrophils, lymphocytes, monocytes, eosinophils, and basophils. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Groups:
- OLE Period: Placebo/Tolebrutinib: Participants who completed the DB period entered the OLE period and received tolebrutinib 60 mg orally once daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 2 | 1
Participants
  Hematocrit | 1 | 0
  Hemoglobin | 1 | 0
  White blood cells | 1 | 0
  Monocytes | 2 | 0

4. Primary Outcome: OLE Period: Number of Participants With Clinical Chemistry Parameter Abnormalities
Description: Clinical chemistry parameters assessed were blood urea nitrogen, creatinine, glucose, total and direct bilirubin, potassium, sodium, chloride, bicarbonate, calcium, albumin, creatine phosphokinase, alkaline phosphatase, aspartate aminotransferase/serum glutamic-oxaloacetic transaminase, alanine aminotransferase/serum glutamic-pyruvic transaminase, lipase, and total protein. Only the category (Alkaline phosphatase) in which at least 1 participant had data were reported.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 2 | 1
Participants | 0 | 1

5. Primary Outcome: OLE Period: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: ECG parameters assessed were heart rate, pulse rate, QRS interval, QT interval and QT interval corrected using Fridericia's formula [QTcF]).
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

6. Primary Outcome: OLE Period: Number of Participants With Vital Signs Abnormalities
Description: Vital signs assessed were heart rate, systolic blood pressure, diastolic blood pressure, weight and temperature. Only those category (Weight >=5% decrease from Baseline) in which at least 1 participant had data were reported.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: Analysis was performed on the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 2 | 1
Participants | 1 | 0

7. Secondary Outcome: DB Period: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Total Score at Week 26
Description: The QMG is a clinician-reported outcome to assess muscle weakness in participants with MG. The QMG test consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item). Each item is scored on 3-point scale ranged from 0 (none) to 3 (severe), where higher score represents most severe muscle weakness. The QMG total score is the sum of each individual item score which ranged from 0 (normal) to 39 (severe). Higher score represents greater disease activity. DB period Baseline value was defined as last available value prior to the first dose of the study medication in the DB period.
Time Frame: Baseline (Day 1), Week 26
Population: as for outcome 1
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: DB Period: Change From Baseline in Quantitative Myasthenia Gravis (QMG) Total Score at Week 12
Description: The QMG is a clinician-reported outcome to assess muscle weakness in participants with MG. The QMG test consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item). Each item is scored on 3-point scale ranged from 0 (none) to 3 (severe), where higher score represents most severe muscle weakness. The QMG total score is the sum of each individual item score which ranged from 0 (normal) to 39 (severe). Higher score represents greater disease activity. The QMG total score at Week 12 is reported in this outcome measure. DB period Baseline value was defined as last available value prior to the first dose of the study medication in the DB period.
Time Frame: Baseline (Day 1), Week 12
Population: Analysis was performed on modified intention-to-treat (mITT) population which included all randomized and treated participants with a Baseline value and at least 1 post-baseline value for any efficacy assessment. Data for this outcome measure was not collected and analyzed for OLE period of the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
score on a scale | -2.0 (7.9) | -1.7 (2.9)

9. Secondary Outcome: DB Period: Change From Baseline in Myasthenia Gravis Impairment Index (MGII) Total Score at Week 26
Description: MGII: measure of MG severity, with demonstrated fatigability, reliability and construct validity. It consists of 22-item patient-reported questionnaire and 6 clinician-assessment items. MGII can be divided into 2 sub-scale-scores: ocular (8 items) & generalized (20 items) impairments. Ocular sub-score: calculated by summing 1 to 6 items from patient questionnaire and items 1 & 2 of clinician-assessment. Generalized score: calculated by adding items 7 to 22 from patient questionnaire & items 3 to 6 from the clinician-assessment. Each item is scored on 4-point scale: from 0 (none) to 3 (severe), where higher score=more disease severity. MGII total score: sum of each item of patient questionnaire (total score:0 [normal] to 23 [severe]) & clinician assessment items (total score:0 [normal] to 61 [severe]); ranged from 0 (normal) to 84 (severe). Higher scores=greater disease severity. DB period Baseline: defined as last available value prior to 1st dose of study medication in the DB period.
Time Frame: Baseline (Day 1), Week 26
Population: as for outcome 1
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: DB Period: Change From Baseline in Myasthenia Gravis-quality of Life 15-item Scale (MG-QoL15) Total Score at Week 26
Description: The MG-QOL15 is a 15-item, participant self-reported QoL instrument for participants with MG. The instrument is developed and validated to evaluate general QoL of participants with MG by a clinician in the practice setting. The domains covered by the questionnaire are mobility (9 items), symptoms (3 items), general contentment (1 item) and emotional well-being (2 items). Each item is scored on a scale of 0 (not at all) to 4 (very much), where higher score indicates severe QoL impairment. The MG-QOL15 total score is the sum of each individual item score and ranged from 0 (none) to 60 (severe). Higher scores indicates greater extent and dissatisfaction with MG-related dysfunction. DB period Baseline value was defined as last available value prior to the first dose of the study medication in the DB period.
Time Frame: Baseline (Day 1), Week 26
Population: as for outcome 1
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: DB Period: Percentage of Participants With Greater Than Equal to (>=) 2-point Improvement (Reduction) in Myasthenia Gravis-activities of Daily Living Total Score at Week 26
Description: The MG-ADL is an 8-item patient-reported categorical scale that assesses MG symptoms and their effects on daily activities. The MG-ADL targeted symptoms and disability across ocular (2 items), bulbar (3 items), respiratory (1 items), and gross motor or limb impairment (2 items) symptoms. It evaluates a participant's capacity to perform different activities in their daily life. Each item is scored on a 4-point scale ranged from 0 (normal) to 3 (severe), where higher score represents the more severe symptoms or impaired performance. MG-ADL total score is the sum of each item score which ranged from 0 (normal) to 24 (severe). Higher score represents severe disability due to MG.
Time Frame: Week 26
Population: as for outcome 1
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: DB Period: Percentage of Participants With >=3-point Improvement (Reduction) in Quantitative Myasthenia Gravis Total Score at Week 26
Description: as for outcome 11
Time Frame: Week 26
Population: as for outcome 1
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: DB Period: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), Adverse Events Leading to Permanent Study Intervention Discontinuation and Adverse Events of Special Interests (AESIs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily have to have a causal relationship with the treatment. A SAEs was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. AESI was defined as one of scientific & medical concern specific to the Sponsor's product or program, for which ongoing monitoring and immediate notification by the Investigator to the Sponsor was considered appropriate. Relatedness to study vaccine was based on Investigator's discretion.
Time Frame: From Day 1 up to Week 26
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
Participants
  AEs | 1 | 2
  SAEs | 1 | 1
  AEs leading to permanent study intervention discontinuation | 0 | 0
  AESIs | 1 | 1

14. Secondary Outcome: DB Period: Number of Participants With Hematological Abnormalities
Description: as for outcome 3
Time Frame: From Day 1 up to Week 26
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
Participants
  Hematocrit | 1 | 1
  Hemoglobin | 1 | 0
  Monocytes | 1 | 0
  Eosinophils | 1 | 0

15. Secondary Outcome: DB Period: Number of Participants With Clinical Chemistry Parameter Abnormalities
Description: Clinical chemistry parameters assessed were blood urea nitrogen, creatinine, glucose, total and direct bilirubin, potassium, sodium, chloride, bicarbonate, calcium, albumin, creatine phosphokinase, alkaline phosphatase, aspartate aminotransferase/serum glutamic-oxaloacetic transaminase, alanine aminotransferase/serum glutamic-pyruvic transaminase, lipase, and total protein. Only those categories in which at least 1 participant had data were reported.
Time Frame: From Day 1 up to Week 26
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
Participants
  Protein | 1 | 1
  Alanine aminotransferase | 1 | 0
  Aspartate aminotransferase | 1 | 0
  Alkaline phosphatase | 0 | 1
  Total bilirubin | 0 | 1

16. Secondary Outcome: DB Period: Number of Participants With Electrocardiogram Abnormalities
Description: ECG parameters assessed were heart rate, pulse rate, QRS interval, QT interval and QTcF.
Time Frame: From Day 1 up to Week 26
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
Participants | 0 | 0

17. Secondary Outcome: DB Period: Number of Participants With Vital Signs Abnormalities
Description: Vital signs assessed were heart rate, systolic blood pressure, diastolic blood pressure, weight and temperature. Only those category (Weight >=5% increase from Baseline) in which at least 1 participant had data were reported.
Time Frame: From Day 1 up to Week 26
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Placebo | DB Period: Tolebrutinib
Number analyzed (Participants) | 3 | 3
Participants | 1 | 0

18. Secondary Outcome: OLE Period: Change From Baseline in Myasthenia Gravis-activities of Daily Living Total Score
Description: The MG-ADL is an 8-item patient-reported categorical scale that assesses MG symptoms and their effects on daily activities. The MG-ADL targeted symptoms and disability across ocular (2 items), bulbar (3 items), respiratory (1 items), and gross motor or limb impairment (2 items) symptoms. It evaluates a participant's capacity to perform different activities in their daily life. Each item is scored on a 4-point scale ranged from 0 (normal) to 3 (severe), where higher score represents the more severe symptoms or impaired performance. MG-ADL total score is the sum of each item score which ranged from 0 (normal) to 24 (severe). Higher score represents severe disability due to MG. OLE period Baseline value was defined as last available value prior to the first dose of the study medication in the OLE period.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: OLE Period: Change From Baseline in Quantitative Myasthenia Gravis Total Score
Description: The QMG is a clinician-reported outcome to assess muscle weakness in participants with MG. The QMG test consists of 13 items: ocular (2 items), facial (1 item), bulbar (2 items), gross motor (6 items), axial (1 item), and respiratory (1 item). Each item is scored on 3-point scale ranged from 0 (none) to 3 (severe), where higher score represents most severe muscle weakness. The QMG total score is the sum of each individual item score which ranged from 0 (normal) to 39 (severe). Higher score represents greater disease activity. OLE period Baseline value was defined as last available value prior to the first dose of the study medication in the OLE period.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: OLE Period: Change From Baseline in Myasthenia Gravis Impairment Index Total Score
Description: MGII: measure of MG severity, with demonstrated fatigability, reliability and construct validity. It consists of 22-item patient-reported questionnaire & 6 clinician-assessment items. MGII can be divided into 2 sub-scale-scores: ocular (8 items) & generalized (20 items) impairments. Ocular sub-score: calculated by summing 1 to 6 items from patient questionnaire and items 1 & 2 of clinician-assessment. Generalized score: calculated by adding items 7 to 22 from patient questionnaire & items 3 to 6 from the clinician-assessment. Each item is scored on 4-point scale: from 0 (none) to 3 (severe), where higher score=more disease severity. MGII total score: sum of each item of patient questionnaire (total score:0 [normal] to 23 [severe]) & clinician assessment items (total score:0 [normal] to 61 [severe]); ranged from 0 (normal) to 84 (severe). Higher scores=greater disease severity. OLE period Baseline:defined as last available value prior to 1st dose of study medication in the OLE period.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: OLE Period: Change From Baseline in Myasthenia Gravis-quality of Life 15-item Scale Total Score
Description: The MG-QOL15 is a 15-item, participant self-reported QoL instrument for participants with MG. The instrument is developed and validated to evaluate general QoL of participants with MG by a clinician in the practice setting. The domains covered by the questionnaire are mobility (9 items), symptoms (3 items), general contentment (1 item) and emotional well-being (2 items). Each item is scored on a scale of 0 (not at all) to 4 (very much), where higher score indicates severe QoL impairment. The MG-QOL15 total score is the sum of each individual item score and ranged from 0 (none) to 60 (severe). Higher scores indicate greater extent and dissatisfaction with MG-related dysfunction.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: OLE Period: Percentage of Participants With >=2-point Improvement (Reduction) in Myasthenia Gravis-activities of Daily Living Total Score
Description: as for outcome 18
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: OLE Period: Percentage of Participants With >=3-point Improvement (Reduction) in Quantitative Myasthenia Gravis Total Score
Description: The MG-ADL is an 8-item patient-reported categorical scale that assesses MG symptoms and their effects on daily activities. The MG-ADL targeted symptoms and disability across ocular (2 items), bulbar (3 items), respiratory (1 items), and gross motor or limb impairment (2 items) symptoms. It evaluates a participant's capacity to perform different activities in their daily life, including talking, chewing, swallowing, breathing, brushing their teeth or combing their hair, getting up from a chair, double vision and eyelid droop. Each item is scored on a 4-point scale ranged from 0 (normal) to 3 (severe), where higher score represents the more severe symptoms or impaired performance. MG-ADL total score is the sum of each item score which ranged from 0 to 24, where a higher score represents severe disability due to MG. OLE period Baseline value was defined as last available value prior to the first dose of the study medication in the OLE period.
Time Frame: From Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61)
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: OLE Period: Percentage of Participants Achieving Any Reduction From Baseline of Daily Dose of Oral Corticosteroids (OCS) at Week 61
Description: The use of rescue therapy for generalized MG worsening is allowed at any time during both the DB and OLE parts of the study at discretion of the Investigator in case of at least a 2-point increase of individual non-ocular MG-ADL items compared to the Day 1 MG-ADL value or new or worsening of respiratory/ bulbar symptoms. Rescue therapy includes intravenous immunoglobulin, plasma exchange, change in the standard of care OCS dose or any use of new CS. OLE period Baseline value was defined as last available value prior to the first dose of the study medication in the OLE period.
Time Frame: Baseline (Day 1), Week 61
Population: as for outcome 1
Arm/Group | OLE Period: Placebo/Tolebrutinib | OLE Period: Tolebrutinib/Tolebrutinib
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to Week 26 for DB period and from Week 27 up to Week 61 for OLE period
Description: Analysis was performed on safety population. Based on the low enrolment number and in order to protect and maintain participant privacy/confidentiality, period (DB and OLE) wise data were not reported and only combined analysis was performed.
Groups:
- Placebo: Participants with moderate-to-severe gMG received placebo (matched to tolebrutinib) tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period.
- Tolebrutinib: Participants with moderate-to-severe gMG received tolebrutinib 60 mg tablet orally once daily as an add-on therapy to their SoC for 26 weeks in the DB treatment period. Participants who completed the DB period entered the OLE period and continued to receive tolebrutinib 60 mg orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
  Additionally, participants who received placebo in DB period and completed DB period entered the OLE period and received tolebrutinib 60 mg orally daily along with SoC starting from Week 27 up to an additional 35 weeks in the OLE period until the study termination (i.e., up to Week 61).
Arm/Group | Placebo | Tolebrutinib
All-Cause Mortality (participants affected / at risk) | 0/3 | 1/5
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/5
Other Adverse Events (participants affected / at risk) | 2/3 | 3/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | Tolebrutinib (N=5)
Covid-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=3) | Tolebrutinib (N=5)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 0 (0)
Haemoglobin Decreased (Investigations) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated by the Sponsor due to strategic reasons and was not based on any safety issues. Hence, several planned efficacy analysis were not conducted for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/69/NCT05132569/Prot_SAP_000.pdf